CLINICAL TRIAL: NCT04416360
Title: Clinical Evolution and Parenting in Children and Adolescents With Autism Spectrum Disorder or Attention Deficit Hyperactivity Disorder Quarantined Because of Covid-19 Outbreak
Brief Title: Autism Spectrum Disorder or Attention Deficit Hyperactivity Disorder in Covid-19 Outbreak
Acronym: CLIECO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/20/0151
Record Dates: First submitted 2020-05-19; First posted 2020-06-04 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Autism Spectrum Disorder; Attention-deficit Hyperactivity Disorder
Keywords: home confinement; Covid-19; qualitative research; Autism Spectrum Disorder; Attention-deficit Hyperactivity Disorder
MeSH Terms: conditions — Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Interview by psychologists (Experimental): Children and adolescent interview Parents interview Referring caregiver interview
  Interventions: Other: Interview by psychologists

INTERVENTIONS:
Other: Interview by psychologists — Interviews for children / teenagers and parents :
  * The questions encourage a narrative
  * Repeated interviews: during confinement, at the end of confinement, and 3 months after the end of confinement
  * Interviews carried out by videoconference, by trained psychologists not involved in the care process
  Interview for referring caregivers: a single interview of approximately 45 minutes, 3 months post-confinement

SUMMARY:
In response to the coronavirus disease 2019 (covid-19) outbreak, the home confinement of the population ordered by governments in many countries raise questions about its impact on individuals' physical and mental health in the short and longer term. In children, reduced physical activity, changes in lifestyle, disturbances in sleep patterns, lack of in-person contact with peers, poor or inadequate understanding of health risks may be risk factors of anxiety, stress, fatigue, sleep disorders. These problematic effects could be modulated by social factors (housing in urban or rural areas, availability of personal space at home, parenting stress, etc.).

DETAILED DESCRIPTION:
Children with Autism Spectrum Disorder (ASD) and/or hyperactive children (ADHD) usually have behavioral and emotional difficulties. The disorders they suffer from, which considerably disturb family life, the therapies they benefit from, which help to organize and structure their daily lives, make them a coherent study group whose observation during home confinement is particularly relevant. Therefore, it is especially interesting to explore the impact of quarantine on the evolution of clinical symptoms and family dynamic.

There is little evidence about the impact of prolonged confinement in these children. The first clinical observations, at the beginning of confinement, reported various situations. Some children showed marked emotional disturbances, whereas others seem to be happy with less social pressure. For ASDs, the ritualization can be a stabilizing factor. For ADHDs, the decrease in school pressure is undoubtedly a positive factor. The availability of parents to create a suitable environment could play a major role. In all cases, changes in care management (teleconsultations for most of them), disruption in routines and lack of points of reference, adjustment in parenting and caring for children for the parents (with difficulties that could increase with prolonged duration of confinement), could have serious long-term effects, but also create opportunities.

So, the present study aim to document the experience of home confinement in children and adolescents with ASD and/or ADHD quarantined because of covid-19 outbreak in various socio-cultural contexts. The experiences reported by the children, their parents and their caregivers will help understand the psychological impact of quarantine.

ELIGIBILITY:
1. Inclusion Criteria:

   Children / adolescents:
   * autism spectrum disorder (ASD) w/wo co-morbidities and/or attention-deficit - hyperactivity disorder (ADHD)
   * aged 6 to 17 years (developmental age)
   * cared by child psychiatry services involved in the study with continuing care (teleconsultations) during home confinement
   * at least one parent consent to participate in the study
   * child benefiting from a social security

   Parents: one or both parents depending on availability and confinement configurations (childcare)

   Referring caregivers: the referring caregiver will be identified at the time of the child's inclusion in the study
2. Exclusion Criteria:

   * Parents subject to a judicial safeguard order, guardianship or trusteeship
   * Parents or children/adolescents who refuse to participate
   * Parents unable to comply with the study requirements because of language or because of lack of access to visio or telephone conference facilities

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 35 (Actual)
Dates: Start 2020-05-05 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Interview of the parents : contextual data | Baseline
  composition, home confinement, change in the environment, personal room at home, screens with internet access, parents' current professional status, teleworking, care, family concerns related to Covid-19, parenting stress, schooling, recurrent complaints.
Interview of the children/adolescents/ parents : Experience of the confinement in general | Baseline
  related to education; related to daily family life; related to leisure, related to care (children/adolescents, parents)
Interview of the children/adolescents/ parents : Experience of the confinement in general | 1 month
  related to education; related to daily family life; related to leisure, related to care (children/adolescents, parents)
Interview of the children/adolescents/ parents : Experience of the confinement in general | 3 months
  related to education; related to daily family life; related to leisure, related to care (children/adolescents, parents)
Interview of the referring caregiver : data relating to disease and management of care | 3 months
  Data relating to disease and management of care. Experience of the referring caregiver.

CONTACTS AND LOCATIONS:
Overall Officials: Malika DELOBEL-AYOUB, Principal Investigator — University Hospital, Toulouse
Locations (5):
- France (5):
  - University hospital of Toulouse, Toulouse, Occitanie
  - Centre Hospitalier de Versailles, Le Chesnay
  - Centre Hospitalier Esquirol, Limoges
  - Hôpital Robert-Debré (AP-HP), Paris
  - Maison de Solenn (Hôpital Cochin AP-HP), Paris